CLINICAL TRIAL: NCT00202267
Title: Community Randomised Control Trial of the Effectiveness of Two Compression Bandaging Technologies
Brief Title: Community RCT of the Effectiveness of Two Compression Bandaging Technologies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Margaret Harrison, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCT 63175; 394622
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Venous Ulcer
Keywords: leg ulcer, compression, bandage, APBI, venous insufficiency
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer; Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Clients randomized to short-stretch bandaging application
  Interventions: Device: Short-stretch Bandage (Non-elastomeric)
- 2 (Active Comparator): Clients randomized to four-layer bandaging application
  Interventions: Device: Four-layer Bandage (Elastomeric)

INTERVENTIONS:
Device: Four-layer Bandage (Elastomeric) — Precise components of the four-layer system depend on the circumference of the ankle. All the bandages are discarded after a single use, usually one week.
  Other Names: Profore bandaging system (Smith & Nephew Medical Ltd.)
  Arms: 2
Device: Short-stretch Bandage (Non-elastomeric) — These bandages are applied in a figure-eight technique; two bandages are applied at full extension in opposite directions up the leg (i.e., clockwise and counter clockwise). The participant will wash the short-stretch wherever possible and reused. The number of bandages supplied to each patient will be recorded on the visit record.
  Other Names: Comprilan (Beiersdorf-Jobst, Inc.)
  Arms: 1

SUMMARY:
Leg ulcers are emotionally distressing and painful, and often require months or years to heal. Although rarely acknowledged as a pressing health care issue, leg ulcers comprise a common, complex, and costly condition, managed primarily through community home care services. Indeed, leg ulcers are the most frequently seen and treated chronic wound. There is consensus in recent international, evidence-based practice guidelines that graduated, multi-layer compression is the most effective treatment, and greatly reduces healing time. High compression is more effective than low compression. However, there is no clear evidence as to which high compression technology is the most effective in promoting healing, the most acceptable to patients, or the most cost-effective to the health care system. This study is designed to answer these questions through a randomized trial conducted in the community, where most leg ulcer care currently takes place. Issues such as effectiveness in healing, quality of life, physical discomfort, personal preference, cost to the system and to the individual will be taken into consideration in evaluating two most commonly used types of compression bandaging.

DETAILED DESCRIPTION:
Background:

Although rarely recognized as a pressing health care problem, leg ulcers comprise a common, complex, and costly condition. Over 80% of ongoing management of chronic wounds occurs in the community, and leg ulcers are one of the most frequently seen chronic wounds. The cost of leg ulcer care is considerable, being reported in both the UK and France to account for 2% of their total national health budgets. In Canada, the impact is only now being recognized due to the pressure on home care caseloads resulting from hospital downsizing, nursing shortages, and growing numbers of complex health populations. In one Ontario study, the care for fewer than 200 community leg ulcer cases cost in excess of $1.5 million for supplies and nursing visits, which translates to $100s of millions yearly Canada-wide. The impact on the individual is significant--chronic, painful, and often takes years to heal. Two-thirds of individuals with leg ulcers have at least one recurrence, and 45% have a history with the condition dating back 10 years.

State of Knowledge & Clinical Practice Guidelines:

Over the past decade, evidence from RCT studies and a recent Cochrane systematic review in BMJ demonstrated that venous leg ulcers treated with compression therapy are more likely to heal. Multi-layer high compression systems are more effective than low compression. However, the small number of people in trials comparing different high compression systems meant the review was unable to draw conclusions about their relative merit. Four of these trials have compared 4-layer bandage with short stretch technologies--the most commonly used technologies in Canada. In total, these trials involved only 220 patients, and were thus underpowered. Furthermore, they did not consider factors such as client preference and ease of use, or incorporate an economic evaluation.

Plan of Investigation:

The study will be a multi-centre, pragmatic, randomised trial of two types of compression bandaging technologies, incorporating an economic evaluation.

Research objective: To compare the effectiveness of 2 high compression technologies delivered in the community on ulcer healing, recurrence rates, quality of life, and cost-effectiveness.

Interventions: Four-layer bandage vs. Short-stretch bandage. Sample size: 414 total, 207 in each arm (80% power, " 0.05 to detect 4 week difference in time to heal).

Inclusion Criteria: leg ulcer>1 cm in any one dimension, minimum duration of 1 week, ABPI>0.7.

Randomization: will be carried out and stratified by: Clinical Centre (3 Health Regions in Ontario); Margolis' Prognostic Model (ulcer area and duration), Ulcer episode (1st or recurrent ulcer).

Analysis: Primary outcome: time-to-healing of the reference ulcer.

Secondary outcomes: quality of life & expenditures for treatment. Durability of healing will be assessed-follow-up for up to 52 weeks post-healing to determine recurrence rates associated with both technologies.

Summary:

There is consensus internationally in recommending the application of graduated multi-layer compression. High compression is more effective than low compression; however, there is no clear evidence as to which high compression technology is more effective.

ELIGIBILITY:
Inclusion Criteria:

* clinical presentation of venous insufficiency
* leg ulcer equal to or larger than 0.7 cm in any one dimension
* ulcer a minimum duration of 1 week
* ankle brachial pressure index equal to or greater than 0.80
* participant can provide written consent
* participant can communicate in English, or translation available
* participant 18 years or over

Exclusion Criteria:

* diagnosed with Diabetes Mellitus - insulin dependent or participant on oral hypoglycemics
* participants who failed to improve over a 3-month period after being treated with either the SS or 4-layer compression bandaging system prior to the trial
* previous trial patients (ie individuals previously enrolled in the study but now have recurrence or a new ulcer)
* symptoms of cognitive impairment noted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2004-01; Primary Completion 2008-03 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
4 weeks or greater improvement in time-to-healing with short-stretch bandages compared to the four-layer bandaging system | Time to healing or up to 12 months; post-healing follow-up

SECONDARY OUTCOMES:
rate of reduction in ulcer area | Baseline and time of healing
quality of life | Baseline and every 3 months
expenditures over a one-year follow-up | From baseline to time of healing
Recurrence | Status recorded at last visit of each month; one year post-healing follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Margaret B Harrison, PhD, Principal Investigator — Queen's University; Ian D Graham, PhD, Principal Investigator — University of Ottawa (co-investigator); Elizabeth A Nelson, PhD, Study Director — University of Leeds, UK (co-investigator); Karen Lorimer, MNSc, Study Director — Victorian Order of Nurses (co-investigator); Connie Harris, MNSc, Study Director — ET NOW (co-investigator); Elizabeth VanDenKerkhof, PhD, Study Director — School of Nursing, Queen's University
Locations (15):
- Canada (15):
  - Winnipeg Regional Health Authority, Winnipeg, Manitoba
  - Nursing Practice Solutions, Fort Erie, Ontario
  - VON Hamilton Branch, Hamilton, Ontario
  - Saint Elizabeth Health Care, Kingston, Ontario
  - Kingston Chronic Wound Clinic, Kingston, Ontario
  - ParaMed Health Services, Kingston, Ontario
  - ET Now, Kitchener, Ontario
  - Carefor, Ottawa, Ontario
  - ParaMed Health Services, Ottawa, Ontario
  - St. Joseph's Care Group, Thunder Bay, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - ParaMed Home Health Care, Toronto, Ontario
  - Comcare Health, Toronto, Ontario
  - Ostomy and Wound Care Centre, Regina, Saskatchewan
  - Saskatoon Health Region Home Care, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Vandenkerkhof EG, Hopman WM, Carley ME, Kuhnke JL, Harrison MB. Leg ulcer nursing care in the community: a prospective cohort study of the symptom of pain. BMC Nurs. 2013 Feb 6;12:3. doi: 10.1186/1472-6955-12-3. PMID 23388350
- [Derived] Pham B, Harrison MB, Chen MH, Carley ME; Canadian Bandaging Trial Group. Cost-effectiveness of compression technologies for evidence-informed leg ulcer care: results from the Canadian Bandaging Trial. BMC Health Serv Res. 2012 Oct 2;12:346. doi: 10.1186/1472-6963-12-346. PMID 23031428
- [Derived] Harrison MB, Vandenkerkhof EG, Hopman WM, Graham ID, Carley ME, Nelson EA; Canadian Bandaging Trial Group. The Canadian Bandaging Trial: Evidence-informed leg ulcer care and the effectiveness of two compression technologies. BMC Nurs. 2011 Oct 13;10:20. doi: 10.1186/1472-6955-10-20. PMID 21995267
- See also: Canadian Institutes of Health Research — http://www.cihr-irsc.gc.ca/